CLINICAL TRIAL: NCT06838767
Title: Effectiveness of Kinetic Chain Approach for Rotator Cuff Tendinopathy
Brief Title: Kinetic Chain Approach for Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/02004 Tayyaba Jabeen
Record Dates: First submitted 2024-11-25; First posted 2025-02-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Rotator cuff injury; kinetic chain approach; pain; functional disability; kinesiophobia
MeSH Terms: conditions — Rotator Cuff Injuries; Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinetic chain approach (Experimental): Kinetic chain approach Shoulder flexion with ipsilateral anterior step-up, Shoulder-dump exercise Starting position with Body weight is on the contralateral-side leg with trunk flexion and rotation. Finishing position. With Body weight is on the ipsilateral-side leg with thoracic extension. Modified shoulder-dump Exercise Sternal-lift starting position with head and trunk flexed forward. Finishing position with emphasizing thoracic extension. Tubing fencing exercise starting position with body weight on the ipsilateral leg. Elbow is at the hip; thoracic extension and scapular retraction are encouraged, Athletic stance during ball-stabilization exercise. Axially loaded wall-slide exercise. Motion at the hips and trunk complements the sliding pattern of the hand.Perform each exercise for 3 Days (twice a day) a week for 6 weeks. 10 reps ,2 sets According to FITT protocol, 10 reps, two sessions per day, and three days per week for 6 consecutive weeks.
  Interventions: Other: Kinetic chain approach
- conventional treatment (Active Comparator): 10 min moist heat pack Self-assisted anterior capsular stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Self-assisted posterior capsular stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Self -assisted inferior capsule stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Codman's pendular exercises 10 reps Muscle strengthening exercises (after 4 weeks)
  * Internal rotators and External rotators isometrics Hold for 5-8 seconds and repeat 10 times
  * chair press According to FIIT protocol 10 reps progressing to 20 and 30 repetitions in 5th and 6th week with two session in a day, three days per week for six consecutive weeks
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Conventional treatment — 10 min moist heat pack Self-assisted anterior capsular stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Self-assisted posterior capsular stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Self -assisted inferior capsule stretching Hold for 30 sec and repeat 5 times with 10 sec rest between each stretch Codman's pendular exercises 10 reps Muscle strengthening exercises (after 4 weeks)
  * Internal rotators and External rotators isometrics Hold for 5-8 seconds and repeat 10 times
  * chair press According to FIIT protocol 10 reps progressing to 20 and 30 repetitions in 5th and 6th week with two session in a day, three days per week for six consecutive weeks
  Arms: conventional treatment
Other: Kinetic chain approach — Kinetic chain approach Shoulder flexion with ipsilateral anterior step-up, Shoulder-dump exercise Starting position with Body weight is on the contralateral-side leg with trunk flexion and rotation. Finishing position. With Body weight is on the ipsilateral-side leg with thoracic extension. Modified shoulder-dump Exercise Sternal-lift starting position with head and trunk flexed forward. Finishing position with emphasizing thoracic extension. Tubing fencing exercise starting position with body weight on the ipsilateral leg. Elbow is at the hip; thoracic extension and scapular retraction are encouraged, Athletic stance during ball-stabilization exercise. Axially loaded wall-slide exercise. Motion at the hips and trunk complements the sliding pattern of the hand.Perform each exercise for 3 Days (twice a day) a week for 6 weeks. 10 reps ,2 sets According to FITT protocol, 10 reps, two sessions per day, and three days per week for 6 consecutive weeks.
  Arms: Kinetic chain approach

SUMMARY:
The aim of this research is to determine the effectiveness of the kinetic chain approach on pain, functional disability and kinesiophobia in patient with rotator cuff tendinopathy. Randomized controlled trials done at National institute of rehabilitation and medicine. The sample size was 44. The subjects were divided in two groups, 22 subjects in Group A that received Conventional Treatment and 22 subjects in Group B that received Kinetic chain approach and conventional treatment. Study duration was of 6 months. Sampling technique applied was non probability connivance sampling technique. Patient with age between 40 to 65 years, Clinically diagnosed and Patients who meet the diagnostic criteria ≥ three positives in five shoulder impingement tests: Neer's sign, Hawkins and Kennedy test, Empty Can test, painful arc of abduction, and external rotation (ER) resistance test, Patients in acute (4 weeks) and sub-acute stage (4-6 weeks).Patients with positive scapular assistance test (SAT) and scapular retraction test (SRT). Were included. Tools used in the study are NPRS (Numeric Pain Rating Scale). SPADI (Shoulder Pain and Disability) .Tampa Scale for Kinesiophobia TSK-11. Data was be analyzed through SPSS -25

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Age between 40 to 65 years.
* Clinically diagnosed and Patients who meet the diagnostic criteria ≥ three positives in five shoulder impingement tests: Neer's sign, Hawkins and Kennedy test, Empty Can test, painful arc of abduction, and external rotation (ER) resistance test (14)
* Patients in acute (4 weeks) and sub-acute stage (4-6 weeks).
* Patients with positive scapular assistance test (SAT) and scapular retraction test (SRT).

Exclusion Criteria:

* Patients with Cervical radiculopathy or previous shoulder surgery.

  * Any Participants with a full thickness tear of rotator cuff tendon.
  * History of glenohumeral dislocation, or other traumatic injury to the shoulder
  * Diagnosed patients of rheumatoid arthritis and osteoarthritis.
  * Hemiplegia affecting the shoulder and lower extremity
  * A complex myofascial pain syndrome.
  * History of significant lower extremity problems, including severe joint pain, recent fractures, or major musculoskeletal disorders (e.g. chronic ligament injuries)

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
NPRS (Numeric Pain Rating Scale) | 6 weeks
  NPRS (Numeric Pain Rating Scale) the NPRS is an 11-point ordinal system, used measure subject perceived level of pain .Assess pain intensity at baseline, 9 session and after 18 session

SECONDARY OUTCOMES:
SPADI (Shoulder Pain and Disability Index) | 6 weeks
  SPADI (Shoulder Pain and Disability Index) is a patient completed questionnaire with 13 items. The pain subscale has 5-items and the Disability subscale has 8-items. Assess outcome at baseline , 9th session and after 18 session
Tampa Scale for Kinesiophobia TSK-11 | 6 weeks
  Tampa Scale for Kinesiophobia TSK-11 Originally 17 item scale, used to identify fear or movement or re-injury. Assess outcome at baseline, after 9th session and after 18th session

CONTACTS AND LOCATIONS:
Overall Officials: Aneela Zia, MsOMPT, Principal Investigator — Riphah International University
Locations (1):
- National institute of rehabilitation medicine , polyclinic islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No